CLINICAL TRIAL: NCT04285489
Title: A Multi-center, Retrospective Registry Study on the Safety of Hakim Programmable Shunt System
Brief Title: A Study on the Safety of Hakim Programmable Shunt System
Status: Completed | Type: Observational
Sponsor: Integra LifeSciences Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: C-HAKIM-001
Record Dates: First submitted 2020-02-24; First posted 2020-02-26 (Actual); Results first posted 2021-09-21 (Actual); Last update posted 2021-11-05 (Actual); Status verified 2021-11

CONDITIONS: Hydrocephalus
MeSH Terms: conditions — Hydrocephalus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Hakim Shunt Programmable System — patient accept Hakim Shunt Programmable System due to HCP

SUMMARY:
This study aimed to collect safety information from subjects implanted with a shunt system (trade name: Hakim Shunt Programmable System) produced by Codman & Shurtleff, Inc. of the United States. Device safety would be assessed based on all the adverse events that occurred within one year after the subjects implanted the catheter.

ELIGIBILITY:
Inclusion Criteria:

1. The informed consent was exempted by the Ethics Committee of a research center. Either a subject or his/her legal representative signed the informed consent form (ICF) prior to enrollment.
2. Subject had an indication suitable to use Hakim Shunt Programmable System.
3. Subject received a Hakim Shunt Programmable System at least one year ago.

Exclusion Criteria:

1. Subject didn't have an indication suitable to use the product.
2. Subject was known to be allergic to a component or ingredient of the product to be implanted, including silicone tubing and other components.
3. According to the comprehensive judgment of an investigator, subject had an infection of the implant site when the shunt system was implanted, such as ventriculitis, meningitis, peritonitis, and local implant skin infection.
4. Subject was simultaneously implanted with another shunt system different from Hakim Shunt Programmable System.
5. Subject had a contraindication of the shunt operation.
6. Subject had uncorrected coagulopathy or any bleeding disorder.

Ages: 2 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with an implanted Hakim catheter due to Hydrocephalus (HCP)
Sampling Method: Non-Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2020-05-02 (Actual); Primary Completion 2020-07-28 (Actual); Study Completion 2020-07-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hua Tang, MD, Study Director — Integra LifeSciences Corporation
Locations (5):
- China (5):
  - Xuanwu Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Guangzhou Women and Children Medical Center, Guangzhou, Guangdong
  - Tongji Hospital of Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Nanjing Brain Hospital Affiliated to Nanjing Medical University, Nanjing, Jiangsu
  - West China Hospital of Sichuan University, Chengdu, Sichuan

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in Xuanwu Hospital, Capital Medical University, Guangzhou Women and Children Medical Center, West China Hospital Sichuan University, Tongji Hospital of Tongji Medical College, Huazhong University of Science and Technology, Nanjing Brain Hospital. The first subject was enrolled in May 2, 2020, and all subjects were enrolled before Jul 1, 2020.
Pre-assignment Details: Screened 140 patients, 130 of them were enrolled, including 71 adult patients and 59 minors (subject age below 18). 10 patients were screening failures for inclusion/exclusion criteria deviation.
Groups:
- HAKIM Programmable Shunt System Arm: 130 patients would be enrolled and adverse events would be collected for subjects enrolled within one year after the implantation of HAKIM Programmable Shunt system from April 01, 2017 to August 31, 2019, through case review or hospital database.
Period: Overall Study
Arm/Group | HAKIM Programmable Shunt System Arm
Started (The first subject was enrolled in May 2, 2020) | 130
Completed (all subjects finished the study by Jul 1, 2020.) | 130 (all subjects finished the study before Jul 1, 2020.)
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: 130 enrolled subjects were included into PPS.
Groups:
- HAKIM Programmable Shunt System Arm: One year' safety data of patients implanted HAKIM Programmable Shunt system from April 01, 2017 to August 31, 2019.
Arm/Group | HAKIM Programmable Shunt System Arm
Number analyzed (Participants) | 130
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 59
  Between 18 and 65 years | 71
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.03 (24.48)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54
  Male | 76
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 130
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  China | 130

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Non-infection Within One Year
Description: Non-infection rate of a subject within one year
Time Frame: 1 year
Population: 130 participants implanted Hakim shunting system for 1 year
Measure: Count of Participants; unit: Participants
Groups:
- Treatment Arm, Single Arm Study: This study was designed to be single arm, multi-center, observational and retrospective. It is designed to collect information from actual clinical practice from the clinical records of patients in relation to the one-year clinical safety to the use of operation of HAKIM Programmable Shunt system.
Arm/Group | Treatment Arm, Single Arm Study
Number analyzed (Participants) | 130
Participants | 5

ADVERSE EVENTS:
Time Frame: within 1 year after investigated device implanted
Groups:
- HAKIM Programmable Shunt System Arm: Subject implanted HAKIM Programmable Shunt system for at least of one-year.
Arm/Group | HAKIM Programmable Shunt System Arm
All-Cause Mortality (participants affected / at risk) | 4/130
Serious Adverse Events (participants affected / at risk) | 31/130
Other Adverse Events (participants affected / at risk) | 9/130
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HAKIM Programmable Shunt System Arm (N=130)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Product problems (Product Issues) | 6 (6)
Intracranial infection (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Neurological disorders (Nervous system disorders) | 7 (7)
Injuries (Injury, poisoning and procedural complications) | 6 (6)
Craniosynostosis (Congenital, familial and genetic disorders) | 1 (1)
tumor (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HAKIM Programmable Shunt System Arm (N=130)
Product problems (Product Issues) | 9 (9)
Hyponatremia (Metabolism and nutrition disorders) | 7 (7)
Pneumonia (Infections and infestations) | 9 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-11-18): https://cdn.clinicaltrials.gov/large-docs/89/NCT04285489/Prot_SAP_000.pdf